CLINICAL TRIAL: NCT02462304
Title: To Compare the Efficacy of Monotherapy With Anti-Vascular Endothelial Growth Factor (Ranibizumab or Bevacizumab) Versus Combination Therapy With Anti-Vascular Endothelial Growth Factor and End-point-management Grid Laser Photocoagulation for Diabetic Macular Edema
Brief Title: To Compare Anti-VEGF Monotherapy With Anti-VEGF and EPM Grid Laser Combination Therapy for Diabetic Macular Edema
Acronym: END-DME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The University of Hong Kong (Other)
Collaborators: Nagoya City University (Other); Asahikawa Medical College (Other); University of Fukui (Other); Eguchi Eye Clinic (Other); Kyoto University (Other); Nagasaki University (Other); Osaka Medical College (Other); Kyushu University (Other); Tokyo Medical University Hachioji Medical Centre (Unknown); Hokkaido University (Other); Kyorin University (Other); Inje University (Other); Pusan National University (Other); Kyungpook National University Hospital (Other); Chungnam National University Hospital (Other); Sun Cheon Hyang University (Unknown); Kyunghee University (Other); Yeungnam University Hospital (Other); Korea University (Other); National University Hospital, Singapore (Other); Yamagata University (Other)
Responsible Party: Principal Investigator, Dr. WONG Yat-hin Ian, Clinical Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: END-DME1
Record Dates: First submitted 2015-03-23; First posted 2015-06-04 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Macula Edema
Keywords: Diabetic Macula Edema; End-Point-Management; ranibizumab; bevacizumab
MeSH Terms: interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combination Anti-VEGF and EPM laser (Experimental): Subjects will receive both anti-VEGF injections and EPM laser.
  Interventions: Procedure: End-Point-Management grid laser; Drug: ranibizumab; Drug: Bevacizumab
- Anti-VEGF monotherapy (Active Comparator): Subjects will receive anti-VEGF injections monotherapy.
  Interventions: Drug: ranibizumab; Drug: Bevacizumab

INTERVENTIONS:
Procedure: End-Point-Management grid laser
  Arms: Combination Anti-VEGF and EPM laser
Drug: ranibizumab
Drug: Bevacizumab

SUMMARY:
Objectives:

To compare the efficacy of monotherapy with anti-Vascular Endothelial Growth Factor (ranibizumab or bevacizumab) with combined therapy with anti-Vascular Endothelial Growth Factor and end-point-management grid laser photocoagulation for diabetic macular edema.

Study design:

Open-label non-randomized interventional study.

Study overview:

This study aims to look at the efficacy of treating diabetic macular edema (DME) with either anti-Vascular Endothelial Growth Factor(anti-VEGF) monotherapy, compared with combination therapy with anti-VEGF and End-Point-Management (EPM) grid laser photocoagulation, over a period of 6 months.

Various sites from across Asia (Japan, South Korea, Hong Kong) will participate. Depending on the availability of EPM laser, sites can either contribute to the 'Anti-VEGF monotherapy' arm, or to the 'Combination therapy' arm.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years with CSME
* Diagnosis of diabetes mellitus (type 1 or type 2)
* At least one eye meets the study eye criteria
* Able and willing to provide informed consent prior to any study-related procedures
* Central foveal thickness ≥ 300 microns at baseline (SPECTRALIS or Cirrus HD OCT)
* LogMAR Best corrected visual acuity 0.20 (Snellen 20/30) to 1.3 (Snellen 20/400).
* Willing and able to comply with clinic visits and study-related procedures
* Central Foveal Thickness on OCT 300-600 micron
* After first injection, wait for ME to reduce before proceeding with the laser. Exclude if ME persists >500um at the 4-week follow up

Exclusion Criteria:

* Macular edema is considered to be due to a cause other than diabetic macular edema.
* An ocular condition is present such that, in the opinion of the investigator, visual acuity loss would not improve from resolution of macular edema (e.g., foveal atrophy, VMT, pigment epithelium abnormalities, dense subfoveal hard exudates, non-retinal condition such as glaucoma etc).
* Substantial cataract that, in the opinion of the investigator, is likely to be affecting visual acuity. Likely to be affecting BCVA and performing laser treatment.
* History of treatment for diabetic macular edema at any time in the past (such as grid macular photocoagulation).
* History of treatment for diabetic macular edema at any time in the past 3 months (such as intravitreal or peribulbar corticosteroids, ranibizumab, bevacizumab, aflibercept).
* Focal laser photocoagulation should be performed before enrolling into the study if needed. 3 months gap required between last laser procedure and recruitment.
* History of panretinal (scatter) photocoagulation (PRP) within 3 months prior to enrollment.
* Anticipated need for PRP in the study period.
* History of major retinal surgery (including vitrectomy, scleral buckle, any glaucoma surgery, etc.).
* History of YAG capsulotomy performed within 3 months.
* Aphakia.
* Intraocular pressure ≥ 25 mmHg.
* History of open-angle glaucoma (either primary open-angle glaucoma or other cause of open-angle glaucoma; note: history of angle-closure glaucoma is not an exclusion criterion).
* Exam evidence of external ocular infection, including conjunctivitis, chalazion, or significant Blepharitis.
* Systemic Exclusion Criteria: A subject is not eligible if any of the following exclusion criteria are present:
* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110).
* Major surgery within 28 days prior to randomization or major surgery planned during the next 6 months.
* Myocardial infarction, other cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 6 months prior to randomization.
* Systemic anti-vascular growth factor (ranibizumab) or pro-VEGF treatment within 4 months.
* For women of childbearing potential: pregnant or lactating or intending to become pregnant within the next 12 months.
* Subject is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the study.
* The target eye is the only eye of the subject, with the fellow eye's visual acuity lower than 1.3 LogMAR units.
* Baseline logMAR BCVA from 0.05 to 0.5 (Snellen)
* Fellow eye BCVA 0.05 or worse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Difference in number of anti-VEGF required | 6 months
  The number of injections of anti-VEGF required at the end of the 6 months period.

SECONDARY OUTCOMES:
Change in best corrected visual acuity | 6 months
  The change in best corrected visual acuity among subjects in different groups at the end of the 6 months period when compared to baseline.
Central retinal thickness | 6 months
  The change in central retinal thickness among subjects in different groups at the end of the 6 months period when compared to baseline.
Treatment related complications | 6 months
  This will look at treatment related complications in terms of changes in intraocular pressure post-injection
Treatment related complications | 6 months
  This will look at treatment related complications in terms of infection
Treatment related complications | 6 months
  This will look at treatment related complications in terms of retinal detachment
Recurrence of macular edema | 6 months
  Recurrence of macular edema during the 6 months period will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wong, FRCOphth, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China